CLINICAL TRIAL: NCT06218251
Title: A Prospective, Multi-center, Open-label Study to Evaluate Subject Satisfaction and Natural Outcomes Following Administration of BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex in Subjects With Upper Facial Lines (Glabellar Lines, Lateral Canthal Lines, and Forehead Lines)
Brief Title: A Study to Evaluate Participant Satisfaction and Natural Outcomes Following Administration of BOTOX Cosmetic Injections in Adult Participants for Treatment of Upper Facial Lines
Acronym: UFL BOND 974
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M22-974
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Upper Facial Lines
Keywords: Glabellar Lines; Lateral Canthal Lines; Forehead Lines; BOTOX; Botulinum Toxin Type A; OnabotulinumtoxinA; Upper Facial Lines; Crows Feet Lines; Wrinkles; Facial Wrinkles; Facial Rhytides
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BOTOX (Experimental): Participants will receive injections in the glabellar complex, in each of the lateral canthal area, and in the frontalis muscle on Day 1.
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — Intramuscular Injections
  Other Names: Botulinum Toxin Type A; OnabotulinumtoxinA

SUMMARY:
Facial lines that develop from repeated facial expression, such as glabellar lines (GL), lateral canthal lines (LCL), and forehead lines (FHL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. The purpose of this study is to evaluate participant satisfaction and natural outcomes following the administration of BOTOX Cosmetic in adult participants with upper facial lines (GL, LCL, and FHL).

This is an open-label study in which all participants will receive active study treatment. Around 100 adult participants with an assessment of moderate to severe GL, LCL, and FHL, will be enrolled at approximately 10 sites in the United States and Canada.

Participants will receive BOTOX Cosmetic as intramuscular injections to the glabellar lines, lateral canthal lines, and forehead lines at Day 1.

Participants will attend regular visits during the study. The effect of the treatment will be checked by medical assessments for side effects and questionnaires will be completed during regular study visits.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Glabellar Lines, Lateral Canthal Lines, and Forehead Lines.
* Sufficient visual acuity without the use of eyeglasses (contact lens use acceptable) to accurately assess their facial wrinkles.

Exclusion Criteria:

* Presence or history of any medical condition that may place the participant at increased risk to BOTOX Cosmetic or interfere with the study evaluation.
* Presence of tattoos, jewelry, or clothing which obscures or interferes with the target area of interest and cannot be removed.
* History of known immunization or hypersensitivity to any botulinum toxin serotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (7):
  - Skin Wellness Dermatology - Homewood /ID# 248469, Birmingham, Alabama
  - The Research Center at The Maas Clinic /ID# 256633, San Francisco, California
  - Pacific Clinical Innovations /ID# 248467, Vista, California
  - Kavali Plastic Surgery and Skin Renewal Center /ID# 248472, Atlanta, Georgia
  - Tennessee Clinical Research Center /ID# 259161, Nashville, Tennessee
  - Integrated Aesthetics - Spring /ID# 257738, Spring, Texas
  - SkinDC /ID# 248470, Arlington, Virginia
- Canada (3):
  - Skin Matters Medical Aesthetic Centre /ID# 249539, Vancouver, British Columbia
  - Project Skin MD - Ottawa /ID# 249718, Ottawa, Ontario
  - Bertucci MedSpa Inc. /ID# 249757, Woodbridge, Ontario

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-974

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOTOX
Started | 100
Completed | 96
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat Population
Arm/Group | BOTOX
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 66
  More than one race | 5
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Responder Status of 'Mostly Satisfied' or 'Very Satisfied' on the Facial Line Satisfaction Questionnaire (FLSQ) Follow Up Item 4 (Satisfaction With the Natural Look)
Description: The FLSQ consists of 13 questions that assess treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with upper facial lines using the FLSQ 5-point scale where: -2=Very dissatisfied and 2=Very satisfied.
Time Frame: Day 30
Population: Modified Intent-to-Treat Population
  N is Number of subjects with observed measurements at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | BOTOX
Number analyzed (Participants) | 95
Participants | 86

2. Secondary Outcome: Change From Baseline in Overall Score of the Participant's Assessment of FACE-Q Psychological Function
Description: The FACE-Q Psychological Function is a 10-item scale that measures psychological function. The responses score ranges from 0 to 100. Higher scores reflect a better outcome.
Time Frame: Day 30
Population: Modified Intent-to-Treat Population
  N is Number of participants with observed measurements at both baseline and the given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BOTOX
Number analyzed (Participants) | 83
units on a scale | 20.1 (17.96)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 182 days for BOTOX.
Arm/Group | BOTOX
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 19/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOTOX (N=100)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1)
FACIAL DISCOMFORT (General disorders) | 2 (2)
BRONCHITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
DYSPLASTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEADACHE (Nervous system disorders) | 6 (9)
BROW PTOSIS (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT06218251/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT06218251/SAP_001.pdf